CLINICAL TRIAL: NCT05831787
Title: Monitoring SARS-CoV-2 Vaccines and COVID-19 Related Outcomes in Individuals With Multiple Myeloma
Brief Title: COVID19 OutcomeS in Myeloma and the Impact of VaCcines
Acronym: COSMIC
Status: Active, not recruiting | Type: Observational
Sponsor: ASH Research Collaborative (Other)
Collaborators: ModernaTX, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: ASH RC DH 2022-00001
Record Dates: First submitted 2023-04-20; First posted 2023-04-26 (Actual); Last update posted 2024-06-17 (Actual); Status verified 2024-06

CONDITIONS: Multiple Myeloma
Keywords: Myeloma; COVID-19; Vaccine; COSMIC
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell; COVID-19 | interventions — Patient Reported Outcome Measures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Diagnosis of multiple myeloma and currently receiving active treatment for any phase of the disease: Diagnosis of multiple myeloma must meet the International Myeloma Working Group criteria.
  Interventions: Other: Patient Reported Outcomes

INTERVENTIONS:
Other: Patient Reported Outcomes — Patients will be asked to complete baseline, 30-day, and 6-month clinical and patient reported outcome health surveys.

SUMMARY:
The COVID-19 pandemic has had an outsized impact on individuals with underlying social and medical vulnerability, leading to increased rates of severe disease, hospitalization, and death in these groups. Participants with underlying immune compromise, such as those with multiple myeloma, represent one such group. The advent of vaccines against SARS-CoV-2 has significantly limited morbidity and mortality across all groups, but the effectiveness of vaccination in individuals who are less likely to mount sufficient antibody response is uncertain. For this reason, booster vaccines have been recommended for those with underlying immune compromise. However, several key gaps remain in our understanding of how to best protect these individuals.

There is a dearth of real-world evidence about the effectiveness of vaccination and boosters in patients who are immunocompromised, and very little information specifically about the recently approved mRNA boosters. Additionally, rates of vaccination and booster uptake in the United States remain low. A rapid, decentralized method of ascertaining information related to booster vaccine response and adverse events related to vaccines and COVID-19 infection is critical not only to answer questions about the booster vaccines, but to develop an infrastructure for answering similar questions about future vaccines or other diseases.

DETAILED DESCRIPTION:
The purpose of this project is to implement and establish the feasibility of a decentralized real-world evidence study network for patients with multiple myeloma and to monitor outcomes related to COVID-19 infection in this immunosuppressed population. Subjects with multiple myeloma will be invited to participate. The electronic portal will handle all consenting activities. Participants will be asked to complete specific study procedures electronically, including permission for electronic health record (EHR) data transfer. Participants will be asked to complete electronic questionnaires periodically.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of multiple myeloma per the International Myeloma Working Group and currently receiving active treatment for any phase of the disease, including initial therapy, maintenance, or relapsed disease.
* Access to the internet
* An active patient portal (or willingness to activate)
* Willing to electronically sign the study-specific informed consent and authorization form

Exclusion Criteria:

* Non-English speaking
* Lack of internet access
* Cognitive impairment precluding ability to provide informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals with a diagnosis of multiple myeloma per the International Myeloma Working Group and currently receiving active treatment for any phase of the disease, including initial therapy, maintenance, or relapsed disease.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2024-01-23 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility of obtaining baseline clinical and PRO data capture from 200 consented patients. | At Baseline
  Proportion of consented participants who provide responses for the PRO instruments & proportion of participants who permission access to clinical data through the EHR.
Feasibility of obtaining 30-day clinical and PRO data capture from 200 consented patients. | 30 days after enrollment
  Proportion of consented participants who provide responses for the PRO instruments & proportion of participants who permission access to clinical data through the EHR.
Feasibility of obtaining 6-month clinical and PRO data capture from 200 consented patients. | 6 months after enrollment
  proportion of consented participants who provide responses for the PRO instruments & proportion of participants who permission access to clinical data through the EHR.

SECONDARY OUTCOMES:
COVID Vaccine Prevalence | At Baseline
  Percent of patients who enroll on the study platform who had previously received a SARS-CoV-2 booster
COVID Booster Incidence | During 6 month study period
  Percent of patients who enroll on the study platform who went on to receive a SARS-CoV-2 booster after enrollment
PRO Review | During 6 month study period
  Among participants providing PROs, percentage for whom PROs were viewed by site personnel
COVID-19 Infection baseline | At Baseline
  Percentage of participants reporting COVID-19 infection confirmed by home-based or other testing
COVID-19 Infection on study | During 6 month study period
  Percentage of participants reporting COVID-19 infection confirmed by home-based or other testing
Patient reported COVID 19 adverse events baseline | At Baseline
  Patient reported adverse events related to confirmed COVID-19 infection
Patient reported COVID 19 adverse events on study | During 6 month study period
  Patient reported adverse events related to confirmed COVID-19 infection
EHR COVID 19 adverse events baseline | At Baseline
  Hospitalization related to COVID-19 as ascertained by full EHR data transmission provided by permission from the participant
EHR COVID 19 adverse events on study | During 6 month study period
  Hospitalization or death related to COVID-19 as ascertained by full EHR data transmission provided by permission from the participant

CONTACTS AND LOCATIONS:
Overall Officials: William Wood, MD, MPH, Principal Investigator — UNC-Chapel Hill; Saad Usmani, MD,MBA,FACP, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (2):
- United States (2):
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - UNC-Chapel Hill, Chapel Hill, North Carolina

IPD SHARING:
Plan to Share IPD: Undecided
There is no plan at this time. All study data will be stored in the ASH RC Data Hub.

REFERENCES:
- [Derived] Zorger AM, Hirsch C, Baumann M, Feldmann M, Brockelmann PJ, Mellinghoff S, Monsef I, Skoetz N, Kreuzberger N. Vaccines for preventing infections in adults with haematological malignancies. Cochrane Database Syst Rev. 2025 May 21;5(5):CD015530. doi: 10.1002/14651858.CD015530.pub2. PMID 40396505